CLINICAL TRIAL: NCT00799630
Title: Identification of the Effects of NUTRAPERF Consumption on Performance in Endurance-Type Exercise.
Brief Title: Effects of Nutraperf Consumption in Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lescuyer Laboratory (Industry)
Collaborators: Centre Hospitalier Universitaire de Saint Etienne (Other); Université Savoie Mont Blanc (Other)
Responsible Party: Lescuyer laboratory, industry
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 2008-A00982-53
Record Dates: First submitted 2008-11-07; First posted 2008-12-01 (Estimated); Last update posted 2008-12-01 (Estimated); Status verified 2008-11

CONDITIONS: Nutrition Processes
Keywords: energy drink; exercise; BCAA; peripheral and central fatigue
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Carbohydrate drink — Maltodextrins, dextrose, fructose, amino acids (leucine, isoleucine, valine), natural flavors, sodium chloride, magnesium citrate, zinc, lactate, acid: malic acid, anti-caking agent: silicon dioxide; Curcumin (turmeric extract) , Thickener: xanthan gum, caffeine, vitamin C (Acerola extract), vitamin E - B1 - B2 - B3; piperine (black pepper extract).
  Other Names: NUTRAPERF

SUMMARY:
Exercise has numerous health benefits. Nevertheless, when exercise duration is ~45 min or longer and intensity moderate to intense, it may induce different troubles, for example: hypoglycemia, peripheral and central fatigue, muscle damages, osteoarticular injuries, inflammation, cardiovascular dysfunctions. Nutritional loading during exercise may prevent and and/or reduce some of these troubles.

In regard of recent data, we proposed a novel energy drink (NUTRAPERF®) to limit deleterious effects of long time exercise in neutral environment (outside temperature between 4 and 25°C) and to improve performance. If performance may be increased by this energy drink during long time exercise, we proposed that it consumption may also improve performance in short and sub-maximal exercise.

So, the purpose of this study is to investigate the effects of the consumption of this novel energy drink on performance during long and short time exercise. Moreover, we studied the effects of this consumption on different metabolic parameters (heart rate, oxygen consumption, respiratory quotient, ventilation, glycemia, lactatemia), on central and peripheral fatigue and on cognitive parameters.

ELIGIBILITY:
Inclusion criteria

* Man aged between 18 and 45 years.
* Regular sportsman (2 to 4 workouts by week since 3 months minimum).
* Be a long-distance runner.
* Be affiliated or beneficial to the National French Security Social.

Non-inclusion criteria

* Any subject who was injured during the three preceding months study.
* Any subject with a history of disease can disrupt the tests. In particular, subjects with pathological conditions placed on the joints of the knee or ankle (sprain repeated problems or patellar ligament) that could hamper measures of force maximum extension and flexion on these joints or illnesses that prevent the exercise of pedalling or running on treadmill (tendonitis, periostitis) will be excluded.
* Any subject who at the same time participates at another medical experiment.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2008-11

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Physiologie Clinique et de l'Exercice, CHU Saint-Etienne, Saint-Etienne, France

REFERENCES:
- [Derived] Peltier SL, Vincent L, Millet GY, Sirvent P, Morin JB, Guerraz M, Geyssant A, Lescuyer JF, Feasson L, Messonnier L. Effects of carbohydrates-BCAAs-caffeine ingestion on performance and neuromuscular function during a 2-h treadmill run: a randomized, double-blind, cross-over placebo-controlled study. J Int Soc Sports Nutr. 2011 Dec 7;8:22. doi: 10.1186/1550-2783-8-22. PMID 22152427